CLINICAL TRIAL: NCT02131428
Title: Depression and Heart Failure Disease Progression
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00052933
Record Dates: First submitted 2014-04-28; First posted 2014-05-06 (Estimated); Last update posted 2022-01-10 (Actual); Status verified 2021-12

CONDITIONS: Heart Failure
Keywords: Heart Failure; Depression; BNP
MeSH Terms: conditions — Heart Failure; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples with DNA are optional.
Oversight: Data Monitoring Committee: No

SUMMARY:
Heart failure is the most costly diagnosis in the Medicare population. Clinical depression is strikingly common in heart failure patients, and not only diminishes their quality of life, but also is associated with a markedly increased risk of hospitalization or death. This study is designed to further our understanding of the behavioral and biological effects of depression in patients with heart failure, so that appropriate treatments can be developed.

DETAILED DESCRIPTION:
There are over five million Americans living with heart failure (HF), and another 670,000 new cases being diagnosed each year. HF is a characteristically unstable condition that is the most costly diagnosis in the Medicare population and is the most common cause for hospitalization. The instability of HF disease is reflected in short-term fluctuations of the HF disease biomarker, B-Type Natriuretic Peptide (BNP). Patient self-management behaviors are important for minimizing HF disease instability. Depression is often comorbid with HF, and elevated depressive symptoms are associated with a marked increase in adverse clinical outcomes. For both depressed and non-depressed HF patients, worsening depressive symptoms mark a substantially increased risk of cardiovascular hospitalization or death. Despite the risk associated with depressive symptoms, the nature of their association with a worsening HF disease trajectory and adverse clinical outcomes is poorly understood.

Converging evidence suggests that the association between depressive symptoms and accelerated HF disease progression may involve multiple behavioral and pathophysiological pathways. This study proposes an innovative, prospective bio-behavioral monitoring study of 220 HF patients that is designed to address the issue of how depressive symptoms and their bio-behavioral manifestations are implicated in worsening HF disease. Using home-monitoring biotechnology, we propose to track fluctuations in HF disease severity using biweekly assessments of BNP over a 16-week period. Symptoms of depression and HF-related health behaviors also will be assessed biweekly via concurrent monitoring. This biweekly bio-behavioral monitoring will be framed by comprehensive baseline and 4-month assessments of depression, HF disease severity, and pathophysiological mechanisms that have been related to the presence of depressive symptoms and implicated in the progression of HF disease. Clinical outcomes also will be assessed over a 5 year follow-up period. This study will create a unique data structure that will allow us to use contemporary statistical methods that will serve to elucidate causal associations between depressive symptoms, self-management health behaviors, pathophysiological processes, and HF disease progression and clinical outcomes. The study findings are expected to yield important advances in our understanding of why depressive symptoms may be particularly detrimental in the presence of HF and will help to inform the design of future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 21 years or older
* Heart Failure of at least 3-months duration
* Left ventricular Ejection Fraction (EF) ≤ 45% by left ventricular angiography, nuclear wall motion study, or echocardiography, Or
* Preserved ejection fraction with either: Hospitalization within the previous 12 months with management of heart failure as a major component of the care provided; or Elevated natriuretic peptide level (NT-proBNP ≥ 360 pg/ml or BNP ≥ 100 pg/ml) within 6 months of enrollment.
* Undergoing treatment with a stable medication regimen.

Exclusion Criteria:

* Myocardial Infarction (MI), within 1 month of enrollment
* Percutaneous Transluminal Coronary Angioplasty(PTCA), Coronary Artery Bypass Graft (CABG) within 3 month of enrollment
* HF due to correctable cause or condition such as uncorrected primary valvular disease
* Alcohol or drug abuse within 12 months
* Illness such as malignancies that are associated with a life-expectancy of < 12 months
* Current pregnancy
* Inability to provide informed consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women aged 21 years or older with diagnosed heart failure.
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2014-11; Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Time to Hospitalization or Death | 5 years
  Time to hospitalization or death
Change in Quality of Life | Bi-weekly of a 4-month period, 4 months, 1 year
  Psychosocial measures of Quality of Life
Change in Self-Management Behaviors | Bi-weekly of a 4-month period, 4 months, 1 year
  Health Behaviors
Change in Heart Failure Disease Biomarkers | Bi-weekly of a 4-month period, 4 months, 1 year
  Disease Biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Sherwood, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No